CLINICAL TRIAL: NCT03627507
Title: A Randomized Observer-blinded Non Inferiority Trial to Evaluate the Immunogenicity and Safety of Locally Manufactured Hepatitis B Vaccine 'Hepa B' in Bangladeshi Healthy Adults.
Brief Title: Non Inferiority Trial of Locally Manufactured 'Hepa-B' Vaccine in Bangladesh.
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: International Centre for Diarrhoeal Disease Research, Bangladesh (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: PR-18020
Record Dates: First submitted 2018-05-30; First posted 2018-08-13 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2018-05

CONDITIONS: Hepatitis B Infection
Keywords: Hepatitis B, Seroconversion, Seroprotection, Vaccine
MeSH Terms: conditions — Hepatitis B; HIV Seropositivity | interventions — Engerix-B

STUDY DESIGN:
Intervention Model Description: Eligible participants will be assigned to receive the Hepa-B Vaccine and Engerix-B Vaccine, in a 1:1 ratio across the target population according to the randomization schedule. The study agents (Hepa B Vaccine or Engerix B Vaccine) will be labelled as per the randomization list.79 participant will receive locally produced Hepa-B Vaccine and 79 participant of comparator group will receive Engerix B Vaccine.
Who Masked: Investigator, Outcomes Assessor
Masking Description: . Since the test and comparator drugs used in this clinical study have different package of vial, a double blind design is not appropriate. Study investigators along with study staffs involved in safety evaluation and laboratory analysis will be blinded regarding the assigned treatment of the participant. The vaccine administration team will be unblinded to the treatment assignment list. The vaccine administrator team members will not be involved in the evaluation of vaccine safety and laboratory analysis.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hepa B (Experimental): 79 participant will be randomly assigned to the test group for receiving the locally produced 'Hepa-B' vaccine.
  Interventions: Biological: Hepa-B
- Engerix B (Active Comparator): 79 participant will be randomly assigned to the comparator group for receiving 'Engerix-B' vaccine.
  Interventions: Biological: Engerix B

INTERVENTIONS:
Biological: Hepa-B — Incepta will manufacture a locally produced Hepatitis B vaccine named 'Hepa- B' which contain recombinant Hepatitis B surface antigen obtaine. This bulk is formulated to prepare finished dosage to manufacture large scale in fully GMP compliant plant. Incepta has conducted preclinical study at Bioneed, India. After successful completion of preclinical study, this non inferiority clinical trial with innovator product is needed for Licensure in Bangladesh.
  Arms: Hepa B
Biological: Engerix B — .'Engerix B' is a recombinant DNA hepatitis B vaccine. It is sterile suspension of purified surface antigen of hepatitis B virus obtained by culturing genetically yeast cells (Saccharomyces cerevisiae cells), which carry the gene that codes for HBsAg
  Arms: Engerix B

SUMMARY:
Hepatitis B is a common and serious infectious disease of the liver, affecting millions of people throughout the world. Persistent Hepatitis B virus infections may cause development of chronic hepatic insufficiency, cirrhosis and hepatocellular carcinoma. Adding to that, Hepatitis B Virus carriers can transmit the disease for many years. It is transmitted through blood or other body fluids infected with the Hepatitis B virus. It is a major cause of morbidity and mortality in countries like Bangladesh. Immunization with Hepatitis B vaccine has been proved effective to prevent HBV infection. But the vaccines, which are recommended till now, are expensive. Locally manufactured Hepatitis B vaccine will be safe, cost effective and affordable for all.

The test vaccine will induce similar seroprotection rates to hepatitis B one month post-vaccination and at 7 months, one month after the third dose of vaccine compared to reference vaccine. This will be done by comparing the percentages of participants with ≥10 mIU/ml anti-HBs by vaccinated with either Hepa B or Engerix B vaccine. The non-inferiority margin will be 10%.

DETAILED DESCRIPTION:
Research Protocol Title: A randomized observer-blinded non inferiority trial to evaluate the immunogenicity and safety of locally manufactured Hepatitis B Vaccine 'Hepa B' in Bangladeshi healthy adults.

Background (brief):

1. Burden: Hepatitis B is a serious and common infectious disease of the liver, affecting millions of people throughout the world1. The severe pathological consequences of persistent Hepatitis B virus (HBV) infections include the development of chronic hepatic insufficiency, cirrhosis and hepatocellular carcinoma (HCC) 1. More than 2000 million people alive today have been infected with HBV at some time in their lives. 1 Of these, about 350 million remain infected chronically and become carriers of the virus. 1 Three quarters of the world's population live in areas where there are high levels of infection 1. Every year there are over 4 million acute clinical cases of HBV and about 25% of carriers, 1 million people a year, die from chronic active hepatitis, cirrhosis or primary liver cancer 1. HBV prevalence in Bangladesh is 2.3 to 9.7 percent with an approximate carrier pool of 10 million. These include healthy adult population 4.4 to 9.7%, healthy children 3%, school girls 2.3%, a rural community 6.4%, and slum communities 3.8%.2,3 About 25-30% population of Bangladesh do not test positive for HBsAg rather test positive for another marker of HBV that is with anti HBc4. Thus about 50 million Bangladeshi people are infected with HBV and transmission of their blood and body fluids may transmit HBV to healthy uninfected person4.
2. Knowledge gap: The prevention of chronic HBV infection has become a high priority in the global community. Immunization with hepatitis B vaccine is the most effective means of preventing HBV infection and its consequence. Vaccine against hepatitis B was introduced in the early 1980s. Recombinant vaccines became available in the mid 1980s.1 Bangladesh introduced Hepatitis B vaccine in the EPI, immunization schedule in a small scale from 2003 but nationwide it was available from 20095 .The HBV prevalence in Bangladesh is 2.3 to 9.7 percent with an approximate carrier pool of 10 million. These include healthy adult population 4.4 to 9.7%, healthy children 3%, school girls 2.3%, a rural community 6.4%, and slum communities 3.8%2,3 . WHO recommended to vaccinate all children and adolescents younger than 18 years-old living in low or intermediate endemicity and also in these settings to vaccinate people in high-risk groups who may acquire the infection6. Currently there is no locally manufactured Hepatitis B vaccine available in Bangladesh. The results of this study will provide information regarding the immunogenicity and safety of the locally manufactured Hepatitis B vaccine 'Hepa B' as a test vaccine using 'Engerix B' as a comparator vaccine in a non inferiority study design.
3. Relevance: The study of this locally manufactured Hepatitis B vaccine, 'Hepa B' among adults will be able to give us information regarding the safety and immunogenicity of the vaccine and compare this locally produced Hepatitis B vaccine 'Hepa B' with 'Engerix B' vaccine. Hepa B has undergone technology transfer from BioBridge company in Pune, India. Incepta and BioBridge entered into an agreement for transfer of technology for manufacture of locally produced 'Hepa- B' in Bangladesh. The regulatory requirements as well as licensure of the vaccine will be initiated in Bangladesh. Currently there are no locally manufactured Bulk of Hepatitis B available in Bangladesh. Once these clinical trials will be completed, Incepta will apply for licensure of Hepa B to the Bangladesh DGDA. This will significantly reduce the cost of vaccine and ensure availability to the people of Bangladesh. Currently the imported vaccine "Engerix B 1 ml" is sold at a price of 608 taka where as Incepta can sell the product at 500 taka. So, in each unit price difference is 108 taka. As each individual needs 3 doses, so it will be 324 taka saved for each subject. Thus the vaccine cost could be significantly reduced and save a large amount of foreign currency of Bangladesh Government.

   Hypothesis (if any): Locally produced intramuscular non-infectious recombinant DNA vaccine Hepa-B is non inferior in terms of immunogenicity and safety among adults in Bangladesh as compared to Engerix-B.

   Objectives:

   Primary Objective

   • To evaluate and compare the immunogenicity and safety of locally produced Hepatitis B vaccine 'Hepa-B' with Engerix-B among healthy adults in Bangladesh.

   Methods:

   This will be a randomized observer-blinded and comparative study on a total of 158 healthy adult participants. Hepa B (Test group) and Engerix B (Comparator Group) controlled non inferiority study in healthy adult (20-45 years of age). 79 participants will receive Hepa B 1.0 ml and another 79 participants will receive Engerix B 1.0 ml Outcome measures/variables: To evaluate and compare the immunogenicity and safety of locally produced Hepa B with Engerix B.

   Primary Objective:

   • To evaluate and compare the immunogenicity and safety of locally produced Hepatitis B vaccine 'Hepa B' with 'Engerix B' in healthy adults in Bangladesh.

   Primary end points:
   1. The test vaccine will induce similar seroprotection rates to hepatitis B one month post vaccination and at 7 months, one month after the third dose of vaccine compared to comparator vaccine. This will be done by comparing the percentage of participants with ≥10 mIU/ml anti HBs after vaccination with either Hepa B or Engerix B vaccine. The non inferiority margin will be 10%.
   2. Number of immediate reactions reported within 30 minutes after vaccination
   3. Number of solicited adverse events (prelisted in the participant's memory aid) occurring up to 4 days following vaccination.
   4. Number of unsolicited AEs up to 30 days after each dose of vaccination.
   5. Occurrence of serious adverse events (SAEs) throughout the trial.

   Secondary end points:

   1. The Ratio of the GMTs of test and comparator vaccines in different time points.

ELIGIBILITY:
Inclusion Criteria:

1. Considered healthy as per medical judgment of the investigator
2. Age: 20 to 45 years
3. Sex: Male, Female and Transgender
4. For married women, a negative urine pregnancy test (Rapid Diagnostic Test) during screening and prior to first, second and third dose of vaccination.Moreover, medical history will be taken thoroughly by study physician from the woman of childbearing age to completely exclude the probability of pregnancy.The women who are married and living with a partner must agree to use a reliable contraceptive method to prevent pregnancy until final follow-up following vaccination. However abstinence is also acceptable.

Exclusion Criteria:

1. Prior history of hepatitis B infection
2. Vaccination with any hepatitis B vaccine
3. Recent febrile illness (within 2 weeks)
4. Known or suspected hypersensitivity to any component of Hepatitis B vaccine (e.g., aluminium, yeast).
5. History of received hepatitis B immune globulin (HBIG), serum immune globulin, or any other blood-derived product.
6. Known or suspected impairment of immunologic function or recent use of immunomodulatory medications (e.g., systemic corticosteroids) more than 14 days with in last 6 months. Does not include topical and inhaled steroids.
7. Receipt of investigational drugs or other investigational vaccines within 3 months prior to first injection with the study vaccine.
8. Pregnant women, nursing mothers, and women planning to become pregnant within the study period.
9. HBsAg reactive, anti-HBs antibody (≥10mlU/ml), anti-HBc (total) reactive, and abnormal liver function test [serum alanine aminotransferase (ALT) level], serum creatinine and CBC (As mentioned in Appendix IV).

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 158 (Actual)
Dates: Start 2018-07-29 (Actual); Primary Completion 2019-05-27 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
1. The test vaccine will induce similar seroprotection rates at 7 months compared to comparator vaccine. | At 7 months(Study day 210)
  The test vaccine will induce similar seroprotection rates to hepatitis B at 7 months ( study day 210) comparator vaccine.

SECONDARY OUTCOMES:
The Ratio of the GMTs of test and comparator vaccines in different time points. | 30 days after last vaccination
  Comparison of the geometric mean titre among the test and the comparator group.

CONTACTS AND LOCATIONS:
Overall Officials: Firdausi Qadri, PhD, Study Chair — International Centre for Diarrhoeal Disease Research, Bangladesh
Locations (1):
- Mirpur Field Office, Dhaka, Mirpur, Bangladesh

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Mushahwar I. Viral Hepatitis: Molecular Biology, Diagnosis, Epidemiology, and Control. 1st ed. Amsterdam: Elsevier; 2004. Page 31, 79
- [Result] Ghosh, D., Ghosh, C., Nath, M., Safwath, S., Saha, S., & Rowshon, A. (2018). Prevalence of anti-HBc total positivity in an impoverished Urban Community in Banglades. Bangladesh Medical Research Council Bulletin, 43(2), 63-70
- [Result] Ahad M, Alim M. Current Challenges in Hepatitis B. TAJ: The Journal of Teachers Association RMC, Rajshahi. 2006; 19 (1):38-44
- [Result] Mahtab MA, Chaudhury M, Uddin MH, Noor-E Alam SM, Rahim MA, Alam MA, Moben AL, Khondaker FA, Choudhury MF, Sarkar MJ, Poddar PK, Foez SA, Akbar SM. Cost Assessment of Hepatitis B Virus-related Hepatitis in Bangladesh. Euroasian J Hepatogastroenterol. 2016 Jul-Dec;6(2):163-166. doi: 10.5005/jp-journals-10018-1190. Epub 2016 Dec 1. PMID 29201750
- [Result] WHO. EPI Fact Sheet. 2016. http://www.searo.who.int/entity/immunization/data/bangladesh. pdf [Accessed 27 Nov. 2017].
- [Result] WHO. Hepatitis B Fact Sheet. 2017. http://www.who.int/mediacentre/factsheets/fs204/en/ [Accessed 27 Nov. 2017]
- [Result] Bzowej NH. Hepatitis B Therapy in Pregnancy. Curr Hepat Rep. 2010 Nov;9(4):197-204. doi: 10.1007/s11901-010-0059-x. Epub 2010 Sep 9. PMID 20949113
- [Derived] Chowdhury F, Akter A, Rahman Bhuiyan T, Tauheed I, Ahmed T, Ahmmed F, Ahmed F, Karim M, Mainul Ahasan M, Rahman Mia M, Mohammad Ibna Masud M, Wahab Khan A, Masum Billah M, Nahar Z, Khan I, Rahad Hossain M, Ariful Islam AZM, Panday AS, Muktadir Rahman Ashik M, Qadri F. A non-inferiority trial comparing two recombinant vaccines (Hepa-B vs. Engerix-B) for hepatitis B among adults in Dhaka, Bangladesh. Vaccine. 2021 Oct 15;39(43):6385-6390. doi: 10.1016/j.vaccine.2021.09.031. Epub 2021 Sep 22. PMID 34561142